CLINICAL TRIAL: NCT01277237
Title: The Effect Of Omega-3 Fatty Acids on Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Edin2008-008275-34; 2008-008275-34 (EudraCT Number)
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2010-12

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Non alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Omacor; Docosahexaenoic Acids; Fatty Acids, Omega-3; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omacor (Active Comparator)
  Interventions: Drug: Omacor
- Lactose tablet (Placebo Comparator)
  Interventions: Drug: lactose tablet

INTERVENTIONS:
Drug: Omacor — Active comparator: omacor 4g/day
  Other Names: Omega-3; N-3 Fatty acids
  Arms: Omacor
Drug: lactose tablet — placebo: lactose tablet 4g/day
  Other Names: Placebo
  Arms: Lactose tablet

SUMMARY:
There is preliminary evidence that Omega 3, a compound naturally found in fish oil, reduces the amount of fat stored in the liver and improves liver function. The purpose of this study is to see whether this observation is correct.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of non-alcoholic fatty liver disease
* fatty infiltration on ultrasound
* abnormal serum liver function tests.

Exclusion Criteria:

* any other identified cause of chronic liver disease
* the prescription of medication which would cause non-alcoholic fatty liver - disease (e.g. tamoxifen)
* already taking supplementary fish oil
* alcohol intake of >20g/day for women, >40g/ day for men
* known allergy to fish oil
* on anticoagulants (antiplatelets are permitted)
* severe heart failure (NYHA class IV)
* pregnancy/ lactation
* age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Liver appearance on ultrasound | 6 months
  The primary endpoint is improvement in grading on ultrasound assessment at six months. Liver brightness and posterior attenuation on ultrasound has previously been shown to correlate significantly with fat scores on liver biopsy.

SECONDARY OUTCOMES:
Liver function tests | 6 months
  the effect of omega-3 fatty acids on serum liver function tests will be assessed following 6 months of treatment.
hepatocyte mitochondrial function | 6 months
  heptocyte mitochondrial function will be measured by breath testing following 6 months of omega-3 supplementation
Health-related Quality of Life | 6 months
  Health related quality of life scores will be compared with baseline following 6 months of omega-3 supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Hayes, MD PhD, Principal Investigator — Royal Infirmary of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom